CLINICAL TRIAL: NCT01080742
Title: A Prospective Observational Study to Evaluate the Efficacy of Lodoz in a Population of Hypertensive Patients
Brief Title: An Observational Study to Evaluate the Efficacy of Lodoz in a Population of Hypertensive Patients
Acronym: Lodoz OS
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 200006-510
Record Dates: First submitted 2010-03-03; First posted 2010-03-04 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2012-06

CONDITIONS: Hypertension
Keywords: Hypertension; Lodoz; Bisoprolol; Hydrochlorothiazide
MeSH Terms: conditions — Hypertension | interventions — Hydrochlorothiazide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lodoz (Combination of bisoprolol and hydrochlorothiazide) — The investigator will decide in advance the best therapeutic strategy for each subject according to current practice, regardless of the potential participation of this subject in the study.
  Other Names: Lodoz

SUMMARY:
This is an observational, prospective, non-interventional, non-randomised, open label multicentric study planned to be conducted in 1000 subjects with mild to moderate primary hypertension in approximately 20 centres in Thailand. The purpose of this study is to examine the beneficial effects of combination of bisoprolol with hydrochlorothiazide available as Lodoz in treatment of Thai subjects with mild to moderate hypertension. The outcome of the study would also provide information on the optimal daily dosage schedule as well as adherence of Lodoz.

DETAILED DESCRIPTION:
Essential hypertension is a heterogenous multifactorial disease affecting large number of population. Monotherapy treatment in hypertension is often unable to achieve the desired blood pressure (BP) goals and subjects even remain at significant risk for developing cardiovascular disease. The use of combination therapy as first line treatment for hypertension provides a solution to the management problems related to hypertension. Among combination drugs, low dose combinations are useful tools in treating large segments of hypertensive subjects because of their several advantages, such as simplified dosage regimens, improve compliance and hypertensive control, decrease dose dependent side effects as well as reduce costs.

OBJECTIVES

Primary objective:

* To evaluate the efficacy of Lodoz therapy when used in routine clinical practice in subjects with mild to moderate essential hypertension.

Secondary objective:

* To evaluate the discontinuation rate of Lodoz therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Subjects diagnosed with mild to moderate essential hypertension
* Subjects foreseen for Lodoz treatment for hypertension
* Age ≥ 18 years

Exclusion Criteria:

* Subjects treated with Lodoz before study initiation
* Subjects who are pregnant
* Subjects with any known contraindications to Lodoz based on local label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of Thailand diagnosed with mild to moderate essential hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 1007 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Mean systolic blood pressure (SBP) reduction and mean diastolic blood pressure (DBP) reduction at month 3 and 6 from baseline | Baseline and until 6 months of treatment

SECONDARY OUTCOMES:
Response rate for SBP (defined as ≥ 10 mm Hg or SBP < 140 mmHg) | After 3 and 6 months of treatment
Response rate for DBP (defined as ≥ 10 mm Hg or DBP < 90 mmHg) | After 3 and 6 months of treatment
Proportion of subjects having reached target BP level, regarding Thai Hypertension Society guideline | After 3 and 6 months of treatment
  The target BP level according to Thai Hypertension Society guideline is less than 140/90 mm Hg and less than 130/80 mm Hg in those with chronic kidney disease.

CONTACTS AND LOCATIONS:
Overall Officials: Dilok Piyayotai, MD, Principal Investigator — Thammasat Heart Center, Thammasat University Hospital, 95 Moo 1, Klong Nueng, Klong Luang, Pathumthani 12120, Thailand
Locations (1):
- Thammasat Heart Center, Thammasat University Hospital, Pathum Thani, Thailand